CLINICAL TRIAL: NCT01984216
Title: Billroth II Versus Roux-en-Y for the Gastrojejunostomy Reconstruction in the Pancreatoduodenectomy: a Randomized Controlled Study
Brief Title: Billroth II Versus Roux-en-Y for the Gastrojejunostomy in the Pancreatoduodenectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion Miguel Servet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: CIRUGIA-CHN; 2013-000693-30 (EudraCT Number)
Record Dates: First submitted 2013-11-07; First posted 2013-11-14 (Estimated); Last update posted 2016-08-29 (Estimated); Status verified 2016-08

CONDITIONS: Pancreatoduodenectomy
MeSH Terms: interventions — Anastomosis, Roux-en-Y; Gastroenterostomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Roux-en-Y (Experimental): Roux-en-Y for the gastrojejunostomy reconstruction
  Interventions: Procedure: Roux-en-Y for the gastrojejunostomy reconstruction
- Billroth II (Active Comparator): Billroth II for the gastrojejunostomy reconstruction
  Interventions: Procedure: Billroth II for the gastrojejunostomy reconstruction

INTERVENTIONS:
Procedure: Roux-en-Y for the gastrojejunostomy reconstruction
  Arms: Roux-en-Y
Procedure: Billroth II for the gastrojejunostomy reconstruction
  Arms: Billroth II

SUMMARY:
The purpose of this study is to compare the safety and superiority of Roux-Y versus Billroth II gastrojejunostomy reconstruction on delayed gastric emptying after pancreatoduodenectomy.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive series of patients undergoing pancreaticoduodenectomy (PD).
* Given informed consent.

Exclusion Criteria:

* Inability to perform pancreatogastrostomy.
* Resection of other organs, except the superior mesenteric-portal vein.
* Previous gastric surgery.
* Preoperative gastric or duodenal obstruction.
* Previous complex abdominal surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2013-11; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Incidence of delayed gastric emptying (DGE) | 30 day after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Javier Herrera, MD, Principal Investigator — Complejo Hospitalario de Navarra
Locations (1):
- Complejo Hospitalario de Navarra, Pamplona, Navarre, Spain

REFERENCES:
- See also: Navarrabiomed: the biomedical research branch of Complejo Hospitalario de Navarra — http://www.navarrabiomed.es